CLINICAL TRIAL: NCT02989064
Title: Phase 1 Cell Dose Escalation Study to Assess the Safety and Tolerability of Genetically Engineered MAGE-A10ᶜ⁷⁹⁶T in HLA-A2+ Subjects With MAGE-A10 Positive Urothelial, Melanoma or Head and Neck Tumors
Brief Title: MAGE-A10ᶜ⁷⁹⁶T for Urothelial Cancer, Melanoma or Head and Neck Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adaptimmune (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADP-0022-004
Record Dates: First submitted 2016-11-07; First posted 2016-12-12 (Estimated); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Urothelial Carcinoma; Head and Neck Cancer; Melanoma; Bladder Urothelial Carcinoma
Keywords: Cell Therapy; T Cell Therapy; SPEAR T Cell; MAGE-A10; Immuno-oncology; Metastatic; Urothelial Cancer; Previously Treated; T Cell Receptor; Inoperable; Advanced; Cancer; Bladder; Head and neck; Melanoma
MeSH Terms: conditions — Carcinoma, Transitional Cell; Head and Neck Neoplasms; Melanoma; Neoplasm Metastasis; Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Autologous genetically modified MAGE A10ᶜ⁷⁹⁶T cells (Experimental)
  Interventions: Genetic: Autologous genetically modified MAGE A10ᶜ⁷⁹⁶T cells

INTERVENTIONS:
Genetic: Autologous genetically modified MAGE A10ᶜ⁷⁹⁶T cells — Infusion of autologous genetically modified MAGE A10ᶜ⁷⁹⁶T on Day 1

SUMMARY:
This Phase 1 study is designed as a cell dose escalation trial in HLA-A*02:01 and HLA-A*02:06 subjects with MAGE-A10 positive urothelial, melanoma or head and neck tumors. The study will enroll subjects between the ages of 18 and 75 using a modified 3+3 cell dose escalation design, to evaluate dose limiting toxicities and determine the target cell dose range. Following the dose escalation phase, additional subjects will be enrolled at the target cell dose range to further characterize safety and the effects at this cell dose.

The study will take the subject's T cells, which are a natural type of immune cell in the blood, and send them to a laboratory to be modified. The changed T cells used in this study will be the subject's own T cells that have been genetically changed with the aim of attacking and destroying cancer cells. When the MAGE-A10ᶜ⁷⁹⁶T cells are available, subjects will undergo lymphodepleting chemotherapy with cyclophosphamide and fludarabine, followed by T cell infusion. The purpose of this study is to test the safety of genetically changed T cells and find out what effects, if any, they have in subjects with urothelial, melanoma or head and neck cancer.

Subjects will be seen frequently by the Study Physician after receiving their T cells for the next 6 months. After that, subjects will be seen every 3, 6, or 12 months according to the Schedule of Procedures. All subjects completing or withdrawing from the interventional portion of the study will enter a long term follow-up phase for observation of delayed adverse events and overall survival for 15 years post-infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥18 to ≤75 years of age at the time of signing the study informed consent.
2. Subject has histologically confirmed diagnosis of any one of the following cancers: (A) urothelial cancer (transitional cell cancer of the bladder, ureter or renal pelvis), (B) melanoma, or (C) squamous cell carcinoma of the head and neck.
3. Subject is HLA-A*02:01 and/or HLA-A*02:06 positive.
4. Subject has measurable disease according to RECIST v1.1 criteria prior to lymphodepletion
5. Subject meets disease-specific requirements per protocol
6. Subject has anticipated life expectancy > 6 months prior to leukapheresis and >3 months prior to lymphodepletion.
7. Subject's tumor shows positive MAGE-A10 expression
8. Subject has an Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1.
9. Subject has a left ventricular ejection fraction ≥50%.
10. Subject is fit for leukapheresis and has adequate venous access for the cell collection.
11. Female subject of childbearing potential (FCBP) must have a negative urine or serum pregnancy test or male subject must be surgically sterile or agree to use a double barrier contraception method or abstain from heterosexual activity with a female of childbearing potential starting at the first dose of chemotherapy and for 4 months thereafter.
12. Subject must have adequate organ function per protocol

Exclusion Criteria:

1. Subject is HLA-A*02:05 in either allele, HLA-B*15:01 and/or HLA-B*46:01 positive. Subject has any A*02 null allele (designated with an "N", e.g. A*02:32N) as the sole HLA-A*02 allele.
2. Subject has received or plans to receive excluded therapy/treatment prior to leukapheresis or lymphodepleting chemotherapy per protocol
3. Subject that has toxicity from previous anti-cancer therapy must have recovered to ≤ Grade 1 prior to enrollment
4. Subject has history of allergic reactions attributed to compounds of similar chemical or biologic composition to fludarabine, cyclophosphamide or other agents used in the study.
5. Subject had major surgery within 4 weeks prior to lymphodepletion; subjects should have been fully recovered from any surgical related toxicities.
6. Subject has an electrocardiogram (ECG) showing clinically significant abnormality at Screening or showing an average QTc interval ≥450 msec in males and ≥470 msec in females (≥480 msec for subjects with bundle branch block [BBB]) over 3 consecutive ECGs. Either Fridericia's or Bazett's formula may be used to correct the QT interval.
7. Subject has symptomatic CNS metastases.
8. Subject has a history of chronic or recurrent severe autoimmune or immune mediated disease
9. Subject has any other active malignancy besides the tumor under study within 3 years prior to Screening.
10. Subject has uncontrolled intercurrent illness
11. Subject has active infection with HIV, HBV, HCV or HTLV
12. Subject is pregnant or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2020-06-04 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events (AE), including serious adverse events (SAE). | 3 years
  Determine if treatment with autologous genetically modified T cells, (MAGE A10ᶜ⁷⁹⁶T ) is safe and tolerable through laboratory assessments including chemistry, hematology and coagulation; and cardiac assessments, including ECG/troponin.
Evaluation of the persistence of genetically modified T cells | 3 years
  Evaluation of the persistence of the infused T cells in the periphery.
Measurement of RCL in genetically modified T cells. | 3 years
  Evaluation of RCL in Subject PBMCs using PCR-based assay.
Assessment of dose limiting toxicities to determine optimally tolerated dose range | 3 years
  Evaluation of dose limiting toxicities will be performed using the CTCAE Version 4.0
Proportion of subjects with a confirmed Complete Response (CR) and/or Partial Response (PR). | 3 years
  Evaluation of the efficacy of the treatment by assessment of the Overall Response Rate according to RECIST v1.1
Interval between the date of first T cell infusion dose and first documented evidence of CR or PR. | 3 years
  Evaluation of the efficacy of the treatment by assessment of time to first response.
Interval between the date of first documented evidence of CR or PR until first documented disease progression or death due to any cause. | 3 years
  Evaluation of the efficacy of the treatment by assessment of duration of response.
Interval between the date of first documented evidence of SD until first documented disease progression or death due to any cause. | 3 years
  Evaluation of the efficacy of the treatment by assessment of duration of stable disease.
Interval between the date of first T cell infusion and the earliest date of disease progression or death due to any cause | 3 years
  Evaluation of the efficacy of the treatment by assessment of progression-free survival.
Interval between the date of first T cell infusion and date of death due to any cause. | 3 years
  Evaluation of the efficacy of the treatment by assessment of overall survival.
Number and % of subjects having any Long Term Follow Up Adverse Events (AEs) | 15 years post last treatment (infusion)
  * New occurrence of any malignancy
  * New occurrence or exacerbation of a pre-existing neurologic disorder
  * New occurrence or exacerbation of a prior rheumatologic or other autoimmune disorder
  * New occurrence of a hematologic disorder
  * New occurrence of any opportunistic and/or serious infections
  * New occurrence of any unanticipated illness and/or hospitalization deemed related to gene modified cell therapy

CONTACTS AND LOCATIONS:
Overall Officials: David Hong, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (11):
- United States (8):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University - School of Medicine, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Tennessee Oncology - Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt - Ingram Cancer Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- Spain (2):
  - Start Madrid-FJD, Fundación Jimѐnez Díaz, Madrid
  - Hospital Universitario 12 Octubre Avda. de Córdoba, Madrid

REFERENCES:
- [Derived] Hong DS, Butler MO, Pachynski RK, Sullivan R, Kebriaei P, Boross-Harmer S, Ghobadi A, Frigault MJ, Dumbrava EE, Sauer A, Brophy F, Navenot JM, Fayngerts S, Wolchinsky Z, Broad R, Batrakou DG, Wang R, Solis LM, Duose DY, Sanderson JP, Gerry AB, Marks D, Bai J, Norry E, Fracasso PM. Phase 1 Clinical Trial Evaluating the Safety and Anti-Tumor Activity of ADP-A2M10 SPEAR T-Cells in Patients With MAGE-A10+ Head and Neck, Melanoma, or Urothelial Tumors. Front Oncol. 2022 Mar 18;12:818679. doi: 10.3389/fonc.2022.818679. eCollection 2022. PMID 35372008